CLINICAL TRIAL: NCT01316497
Title: Acute Kidney Injury in Children Operated for Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aase and Ejnar Danielsens Foundation (Other); The Augustinus Foundation, Denmark. (Other); Direktør Kurt Bønnelycke and Hustru fru Grethe Bønnelyckes Foundation (Unknown); Helen and Ejnar Bjørnows Foundation (Unknown); Raimond and Dagmar Ringgård-Bohn's Foundation (Other); Grosserer L.F. Foghts Foundation (Unknown); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other); The Dagmar Marshall Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20080052
Record Dates: First submitted 2011-03-10; First posted 2011-03-16 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Ischemic preconditioning; Congenital heart defects; Cardiac surgical procedures; Infant; Child
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (RIPC) (Experimental): See intervention description
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Control (Placebo Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — RIPC was performed by applying a blood pressure cuff around the child's leg. The cuff was inflated to 40 mmHg above the systolic pressure in 4 cycles of 5 minutes. Every cycle of ischemia was followed by 5 minutes of reperfusion. The first RIPC cycle started after anesthesia induction when invasive arterial blood pressure was monitored. Appropriate cuff size was used choosing between four sizes. For reproducibility RIPC was performed on the right leg with only a few exceptions, when the leg was used for invasive catheters.
  Arms: Remote ischemic preconditioning (RIPC)
Procedure: Control — The cuff was applied on the leg without inflation in the control group.
  Arms: Control

SUMMARY:
The purpose of this study was to investigate if repeated inflation of a blood pressure cuff applied around one leg causing mild ischemia ("remote ischemic preconditioning") could protect children operated for congenital heart disease from developing acute kidney injury.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) refers to an intervention of remote, brief ischemia which confers systemic protection against consequences of reperfusion injury in distant organs. RIPC has been shown to protect various organs during major surgeries. Our hypothesis was that RIPC could protect kidney function in children operated for complex congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted for surgery for congenital heart disease

Exclusion Criteria:

* heart surgeries of low complexity such as closure of septal defects, aortico-pulmonary windows, establishment of glenn shunts, subaortic membrane resection, redirection of anomalous pulmonary veins, valvotomies, repair of pulmonary artery stenosis and surgeries without the use of extracorporeal circulation

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | Up to 4 days
  Categorized according to the RIFLE criteria (22): R= risk= increased p-creatinine * 1.5 and/or urine output < 0.5 ml/kg/hour for 6 hours, I= injury= increased p-creatinine * 2 and/or urine output < 0.5 ml/kg/hour for 12 hours, F= failure= increased p-creatinine * 3 or p-creatinine ≥ 350 µmol/L in the setting of an acute increase of at least 44 µmol/L and/or urine output < 0.3 ml/kg/hour for 24 hours or anuria for 12 hours, L= complete loss of renal function for > 4 weeks (need for dialysis for longer than 4 weeks), E= end-stage renal disease (need for dialysis for longer than 3 months).

SECONDARY OUTCOMES:
Arterial blood pressure | Up to 3 days
  Incidence of postoperative low blood pressure (below the age-reference level)
Inotropic Score (IS) | Up to 3 days
  The highest postoperative daily dose (µg/kg//min) was used in the formula: IS = [(dopamine + dobutamine) × 1] + (milrinone × 10) + [(epinephrine + norepinephrine) × 100] to calculate the IS.
Reoperation during hospital stay | 90 days
Length of stay at the ICU | 90 days
Length of hospital stay | 90 days
Mortality | 90 days
  In-hospital mortality
Level of cystatin C in plasma | Up to 4 days
Level of Neutrophil Gelatinase-Associated Lipocalin in plasma and urine | Up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten MR Pedersen, MD, Study Director — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby; Vibeke E Hjortdal, MD PhD DMSc, Principal Investigator — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby; Hanne B Ravn, MD PhD, Study Chair — Department of Anesthesia and Intensive Care, Aarhus University Hospital, Skejby; Johan V Povlsen, MD, Study Chair — Department of Renal Medicine C, Aarhus University Hospital, Skejby; Michael R Schmidt, MD PhD, Study Chair — Aarhus University Hospital; Erland Erlandsen, MSc, Study Chair — Department of Clinical Biochemistry, Viborg Hospital
Locations (1):
- Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Aarhus, Denmark

REFERENCES:
- [Background] Pedersen KR, Povlsen JV, Christensen S, Pedersen J, Hjortholm K, Larsen SH, Hjortdal VE. Risk factors for acute renal failure requiring dialysis after surgery for congenital heart disease in children. Acta Anaesthesiol Scand. 2007 Nov;51(10):1344-9. doi: 10.1111/j.1399-6576.2007.01379.x. PMID 17944638
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696